CLINICAL TRIAL: NCT05049382
Title: Does Extraction Difficulty of Mandibular Impacted Third Molars Mirror Post-op Outcomes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SelcukU01
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Difficulty (Experimental): Classified as low difficulty according to Escoda's classification
  Interventions: Procedure: Extraction of impacted mandibular third molar
- Modarate Difficulty (Experimental): Classified as modarate difficulty according to Escoda's classification
  Interventions: Procedure: Extraction of impacted mandibular third molar
- High Difficulty (Experimental): Classified as high difficulty according to Escoda's classification
  Interventions: Procedure: Extraction of impacted mandibular third molar

INTERVENTIONS:
Procedure: Extraction of impacted mandibular third molar — surgical extraction of impacted mandibular third molar tooth

SUMMARY:
The tooth of the patient who applies to the clinic for the impacted wisdom tooth will be classified according to Escoda's difficulty classification. Before the extraction, patients' interincisal, tragus-commissural, and lateral canthus-angulus distances, Oral Health Impact Profile -14 (OHIP-14) scores, and serum levels of CRP and D-Dimer will be measured.

Operation time will be recorded. After the operation, on 4th-day patients' patients' interincisal, tragus-commissural, and lateral canthus-angulus distances, Oral Health Impact Profile -14 (OHIP-14) scores, and serum levels of CRP and D-Dimer and Visual Analogue Scale (for pain) scores will be measured and recorded. On the 10th day, all these measurements will be repeated.

All recorded data will be evaluated for possible correlations based on extraction difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Having extraction of only the mandibular third molar
* No systemic disease
* Signing an informed consent
* No dental phobia or anxiety
* No lesion around the impacted tooth
* Presence of adjacent second molar

Exclusion Criteria:

* Infection after surgery
* Alveolar osteitis
* Not to participate in any follow-up control appointments

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
interincisal distance change | before the surgery, 4th and 10th days
  The distance between the right upper central incisor incisal line and the right upper incisor incisal line will be measured before the surgery, on the 5th and 10th day. The changes will be evaluated.
tragus-commissura distance | before the surgery, 4th and 10th days
  the distance between tragus and angulus in relevant side will be measured before the surgery, on the 5th and 10th day. The changes will be evaluated.
lateral canthus-angulus distance | before the surgery, 4th and 10th days
  the distance between lateral canthus and angulus in relevant side will be measured before the surgery, on the 5th and 10th day. The changes will be evaluated.
OHIP-14 score | before the surgery, 4th and 10th days
  Oral Health Impact Profile Score(14-70; higher is worse)
VAS score | 4th and 10th days
  Visual analog scale score(0-10; higher is worse)
Operation time | after the operation
  Duration of surgical intervention
CRP serum level | before the surgery and 4th day
  Serum levels of CRP will be measured via blood samples before the surgery and the 5th day.
D-Dimer serum level | before the surgery and 4th day
  Serum levels of D-Dimer will be measured via blood samples before the surgery and the 5th day.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Gürses, Study Chair — Selcuk Universty/Dentistry Faculty; Mert Doğrul, Principal Investigator — Selcuk Universty/Dentistry Faculty
Locations (1):
- Selcuk University, Dentistry Faculty, Selçuklu, Konya, Turkey (Türkiye)